CLINICAL TRIAL: NCT05366244
Title: An Observational, Real World Study to Observe Disease Outcomes in Patients With Mild to Moderate Coronavirus Disease 2019 (COVID-19)
Brief Title: An Observational Study in Patients With Mild to Moderate COVID-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Pudong Hospital (Other)
Collaborators: ShuGuang Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: JT001-010x-COVID-19
Record Dates: First submitted 2022-05-06; First posted 2022-05-09 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: COVID-19
Keywords: Mild to Moderate COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with COVID-19: Mild to moderate COVID-19 patient with at least one risk factor for serve COVID-19 illness or death.

SUMMARY:
The purpose of this study was to observe real-world disease progression in mild-moderate COVID-19 patients with at least one risk factor for serve COVID-19 illness or death.

DETAILED DESCRIPTION:
Screening interested participants should sign the appropriate informed consent (ICF) prior to completion any study procedures.

The investigator will review symptoms, risk factors, and other non-invasive inclusion and exclusion criteria.

The following is the general sequence of events during the 28-day evaluation period:

Completion of baseline procedures Participants were assessed for 28 days and completed all safety monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have a positive SARS-CoV-2 test result.
* Participants who have one or more mild or moderate COVID-19 symptoms.
* Participants who have one or more of the following requirements: ≤7 days from the first positive test for SARS-COV-2 virus infection to Day 1; ≤5 days from the first onset of COVID-19 symptoms to Day 1.
* Participants who satisfy one or more than one of the following high risks for progression to severe COVID-19, including death.
* Participants who understand and agree to comply with planned study procedures.
* Participants or legally authorized representatives can give written informed consent approved by the Ethical Review Board governing the site.
* Capable of giving signed informed consent, including of compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

* Participants who are judged by the investigator as likely to progress to severe/critical COVID-19 prior to randomization.
* Participants who have SpO2≤93% on room air at sea level or PaO2/FiO2≤ 300, or respiratory rate ≥30 per minute.
* Participants who require mechanical ventilation or anticipated impending need for mechanical ventilation.
* Participants who have received or plan to receive a SARS-CoV-2 monoclonal antibody treatment or prevention, or antiviral treatment (including the investigational treatment).
* Participants who have received convalescent COVID-19 plasma treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mild to Moderate COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-05-02 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Time to sustained clinical recovery | Up to 28 days
  Time to sustained clinical recovery

SECONDARY OUTCOMES:
Percentage of the participants who have progression of COVID-19 | Day 1 to 28 days
  Percentage of participants who experience these events: Progress to severe and/or critical COVID-19; Death from any cause
Percentage of participants who experience these events | Day 1 to 28 days
  Percentage of participants who experience these events: Progress to severe and/or critical COVID-19; Death from any cause
Time to sustained disappearance of clinical symptoms | Up to 28 days
  Time to sustained disappearance of clinical symptoms
Percentage of clinical recovery participants | Day 3, 5, 7, 10, 14, 21 and 28
  Percentage of clinical recovery participants from baseline to Day 3, 5, 7, 10, 14, 21 and 28
Percentage of participants with no clinical symptoms | Day 3, 5, 7, 10, 14, 21 and 28
  Percentage of participants with no clinical symptoms from baseline to Day 3, 5, 7, 10, 14, 21 and 28
The change of COVID-19 symptom scores | Day 3, 5, 7, 10, 14, 21 and 28
  The change of "COVID-19 symptom scores" from baseline to Day 3, 5, 7, 10, 14, 21 and 28, the score ranges from 0 to 33 and higher scores mean a worse symptom.
Percentage of participants who turned negative for SARS-CoV-2 | Day 3, 5, 7, 10, 14
  Percentage of participants who turned negative for SARS-COV-2 at Day 3, 5, 7, 10, 14
The change of SARS-COV-2 Ct value | Day 3, 5, 7, 10, 14
  The change of SARS-COV-2 Ct value The change of SARS-COV-2 Ct value at Day 3, 5, 7, 10, 14
Safety assessment Results: such as AEs and SAEs through Day 28 | Up to 28 days
  Safety assessment Results: such as AEs and SAEs through Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Minghua Yu, Principal Investigator — Shanghai Pudong Hospital; Yueqiu Gao, Principal Investigator — ShuGuang Hospital
Locations (2):
- China (2):
  - Shuguang Hospital, Shanghai, Shanghai Municipality
  - Shanghai Pudong Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No